CLINICAL TRIAL: NCT01678989
Title: Evaluation of Brain MRI and Clinical Characteristics of Adolescents With Bipolar Disorder and Children of Parents With Bipolar Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turkish Psychiatry Association (Other)
Responsible Party: Principal Investigator, Seher Akbas, Associate Professor, Turkish Psychiatry Association
Other Study IDs: 4946498
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Children; Cranial MRI
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient group: Children with BD, (20 children) 12-18 year-old who agreed to participate in the study will be established.
- Risk group: Twenty healthy children of 12-18 years old who have mothers and/or fathers who previously assessed by an adult psychiatrist and diagnosed as BD according to DSM-IV diagnostic criteria, and who agreed to participate in the study. The age and gender of the groups will be matched.
- Healthy control group: Twenty participants between the ages of 12-18 who agree to participate in the study and whose family members do not have BD. The age and the gender of the groups will be matched.

SUMMARY:
Genetic transition is important in the etiology of bipolar disorder (BD). So, evaluation of children of BD parents and diagnosed with and BD children whether or not brain has affected zones. These groups were compared to healthy controls and whether or not the mental health of children is influenced will be evaluated by the clinical investigation.

DETAILED DESCRIPTION:
MRI studies in children at risk of BD, our understanding of the neurobiology of BD and abnormalities in the studied regions, regions that predispose to the development of our understanding of PBB will shed light on the etiology of the disorder. In this study, the cranial MRI findings and clinical features in adolescents with bipolar disorder and the same age and sex matched children who have parents with BD and healthy controls were investigated. Since there is few studies that evaluate these three groups, there is a need to increase our knowledge on this issue.

ELIGIBILITY:
Inclusion Criteria:

* Children with BD between the ages of 12-18
* Parents with BD who have children between the ages of 12-18
* Healthy children whose parents do not have BD
* Patients who does not have mental or organic disability to answer the questions
* Graduated from primary school

Exclusion Criteria:

* Patients who have mental or organic disability to answer the questions
* Patients who have a history of any chronic disease which is likely to affect the central nervous system
* Patients who have a contraindication for any first application for Magnetic Resonance Imaging (MRI)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In this study, the cranial MRI findings and clinical features in adolescents with bipolar disorder and the same age and sex matched children who have parents with BD and healthy controls were investigated.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University Medical Faculty Department of Child and Adolescent Psychiatry, Samsun, Turkey (Türkiye)